CLINICAL TRIAL: NCT03826277
Title: The Efficacy of Melanostop Peel in Combination With Specifically Selected Home Care Regimen for Improvement of Melasma
Brief Title: Efficacy of Melanostop Peeling for Improvement of Melasma
Acronym: VIMEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VIST - Faculty of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19/1-SK-KPS
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Melanostop peel treatment group (Experimental): * Adult women aged between 20-50 years old.
  * Melasma on the face
  * Fitzpatrick phototypes I-IV
  * Presenting facial melasma
  * In good health condition
  Interventions: Other: Melanostop peel

INTERVENTIONS:
Other: Melanostop peel — Melanostop peel treatments containing 20% azelaic acid, 10% resorcinol, 6% phytic acid, 3% tranexamic acid. (4 treatments, performed at 2-week intervals), in combination with home care products (twice daily):
  * a facial tonic and cream containing brightening ingredients: vitamin C, niacinamide, alpha arbutin, kojic acid,
  * sunscreen protection cream with SPF 50, protecting against UVA, UVB, HEV and IR

SUMMARY:
Participants with face melasma will receive 4 Melanostop peel treatments containing 20% azelaic acid, 10% resorcinol and 6% phytic acid. Peels will be performed at 2-week interval. They will also receive a facial tonic and cream for at home use, containing brightening ingredients: vitamin C, niacinamide, alpha arbutin, kojic acid. They will also receive sunscreen protection cream with SPF 50, protecting against UVA, UVB, HEV and IR. Products for at home use will be used twice a day, every day. Measurements will be made at baseline, on the day of the forth peel treatment and 4 weeks after the last peel. Measured parameters will be: mMASI score, VisioFace photography analysis, melasma area measurements, and melanin index, ΔE, CIELab colour measurements with Cortex SkinLab Combo (Cortex Technology Asp, Denmark).

ELIGIBILITY:
Inclusion Criteria:

* Adult women aged between 20-50 years old.
* Melasma on the face
* Fitzpatrick phototypes I-IV
* Presenting facial melasma
* In good health condition

Exclusion Criteria:

* Breastfeeding and pregnancy
* Women presenting oral herpes
* Other skin diseases, arthritis, diabetes, diseases of thyroid gland
* Any known allergies to ingredients of the products used in the study
* Systemic or topical use of corticosteroids in the previous 6 months
* Antiaging or lightening cosmetic/estetic procedures in the last 2 months (for example: laser or IPL treatments, chemical peels,..)
* Taking drugs for skin lightening in the previous 2 months
* Smoking
* Lesions of unknown origin
* Oral or topical use of isotretinoin in the previous 6 months
* Active bacterial, viral or fungal infections of the skin
* Presence of keloid scars
* Immunodeficiency
* Moderate to severe acne
* Planned change in hormonal contraception or taking drugs that have an affect on hormonal balance during the course of the study
* Unrealistic expectations
* Refusal to use sunscreen protection and complying with instructions

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women
Enrollment: 10 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Modified Melasma Area and Severity Index (mMASI) | week 1, week 7, week 11
  Melasma severity will be evaluated according to Modified Melasma Area and Severity Index (mMASI). Significant change of the mMASI score from baseline is expected bfore 4th and one month after 4th Melanostop peel treatments.
  mMASI score is calculated by first assesing the hyperpigmented area of the face. Four areas are evaluated: forehead (F), right malar region (RM), left malar region(LM), and chin (C), corresponding to 30%, 30%, 30% and 10% of the total face. The melasma in each of the four areas is given a numerical value by rating darkness (D) and area of involvement (A).
  Scoring system: Area of involvement (A), rated 0 to 6: 0= absent; 1 = <10%; 2 = 10% to 29%; 3 = 30% to 49%; 4= 50% to 69%; 5= 70% to 89%; 6= 90% to 100%. Darkness (D), rated 0 to 4: 0= absent; 1= slight; 2= mild; 3= marked; 4= severe.
  mMASI total score = (0,3 x A(F) x D(F) ) + (0,3 x A(LM) x D(LM)) + (0,3 x A(RM) x D(RM)) + (0,1 x A(C) x D(C))
  Total mMASI score range: 0 - 24
Colour difference | week 1, week 7, week 11
  CIE Lab colour will be measured within the lesion and on the control area outside of the lesion using Cortex Dermalab Combo and colour difference (delta E) will be calculated between the areas and in comparison to baseline values.
  Significant change of the melasma colour from baseline and in comparison to control area is expected after 4 Melanostop peel treatments.
Melanin index change | week 1, week 7, week 11
  Melanin index will be measured within the lesion and on the control area outside of the lesion using Cortex Dermalab Combo Skin colour probe. Melanin index is given on a scale 0.0-99.9.
  Significant change of the melanin index from baseline and in comparison to control area is expected before 4th Melanostop peel treatments and 4 weeks after last treatment.
Area of the melasma | week 1, week 7, week 11
  Melasma area will be measured using Visioface photography analysis. Significant change of the melasma area from baseline is expected before 4th Melanostop peel treatments and 4 weeks after last treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Katja Žmitek, PhD, Study Chair — Head of Reasearch Group
Locations (1):
- Higher School of Applied Sciences, Institute of Cosmetics, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No